CLINICAL TRIAL: NCT02683954
Title: The Association Bet Endometriosis, Obesity and nesfatin1
Brief Title: The Association Between Endometriosis, Obesity and nesfatin1
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: nesfatin 1
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- endometriosis: 30 women with laparoscopically diagnosed endometriosis. This group will be categorized into 3 sub-groups according to the BMI: i) Lean: BMI <25.0 kg/m2. ii) Overweight: BMI ≥25.0 kg/m2 but less than 30 kg/m2. iii) Obese: BMI ≥30 kg/m2.
- control: 30 women without any laparoscopically detected pelvic endometriotic pathology. This group will be categorized into 3 sub-groups according to the BMI: i) Lean: BMI <25.0 kg/m2. ii) Overweight: BMI ≥25.0 kg/m2 but less than 30 kg/m2. iii) Obese: BMI ≥30 kg/m2.

SUMMARY:
The association between endometriosis, obesity and nesfatin1.

DETAILED DESCRIPTION:
All women in this study were subjected to all of the following:

1. Verbal consent was obtained.
2. History taking:

   1. Personal history.
   2. Menstrual history.
   3. Use of contraception.
   4. Use of any hormonal treatment in the three months prior to the laparoscopy.
   5. History of infertility and its duration and type.
   6. Sexual history.
   7. Past history.
3. Complete physical examination: general, abdominal and local gynecological examination.
4. Complete preoperative workout for laparoscopy was done.
5. Laparoscopy was done postmenstrual, during follicular phase. All patients gave an informed consent and were fasting for at least 8 hours prior to the laparoscopy, and general anesthesia was used for all patients.

   The pelvis and its structures were observed and checked for presence of endometriotic lesions (uterus, tubes, ovaries and ovarian fossae, uterosacral ligaments, Douglas pouch, uterovesical pouch, broad ligaments and lateral pelvic walls).

   The Endometriotic patients were then classified into stages I-IV according to the revised American Fertility Society scoring system for endometriosis.
6. Venous samples for measurement of nesfatin-1 were taken by venipuncture from patients during the laparoscopy procedure immediately after initial evaluation and before any intervention.
7. Biopsy from lesions suspected as endometriosis was taken during laparoscopy and sent to histopathology for confirmation.
8. The blood samples were centrifuged immediately after their collection at 5000 rpm for 10 min and serum samples were stored at -20 °C until analysis.

   Patients and Methods

   -67-
9. Nesfatin-1 was measured by Enzyme-Linked Immuno Sorbent Assay "ELISA" technique using commercially available kits (Boster Biological Technology Human Nesfatin-1 ELISA kits, Catalog number EK1138, USA) in the Central Labs of Ain Shams University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age group scheduled for laparoscopy for any indication.

Exclusion Criteria:

* Women subject to any hormonal therapy in the last 3 months.
* Women with chronic endocrine disease like diabetes mellitus.
* Women diagnosed with pelvic inflammatory disease (PID).
* Severe medical disorder that prohibits the laparoscopic procedure, such as cardiovascular disease and pulmonary disease.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: sixty female patients were admitted to the wards to undergo laparoscopy for various indications
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Ain Shams University Maternity Hospital, during the period from December 2014 till October 2015. After approval of the research and ethics committee and, sixty patients were admitted to the wards to undergo laparoscopy for various indications and were included in this study.
Period: Overall Study
Arm/Group | Endometriosis | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: sixty patients were admitted to the wards to undergo laparoscopy for various indications and were included in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometriosis | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.83 (3.89) | 29.06 (4.25) | 27.95 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
weight [Mean (Standard Deviation); unit: kilograms] | 66.36 (6.04) | 76.31 (8.35) | 71.34 (8.80)
height [Mean (Standard Deviation); unit: centimeters] | 161.73 (3.99) | 161.16 (4.33) | 161.45 (4.14)
body mass index [Mean (Standard Deviation); unit: kilograms per squared meter] | 25.4 (1.90) | 29.4 (2.86) | 27.4 (3.14)
parity [Number; unit: participants]
  para 0 | 20 | 13 | 33
  para 1 | 10 | 7 | 17
  para 2 | 0 | 8 | 8
  para 3 | 0 | 2 | 2
number of abortions [Number; unit: participants]
  no abortions | 25 | 25 | 50
  one abortion | 4 | 5 | 9
  two abortions | 0 | 0 | 0
  three abortions | 1 | 0 | 1
previous ectopic pregnancies [Number; unit: participants]
  no ectopic | 29 | 28 | 57
  previous ectopic | 1 | 2 | 3
number of living children [Number; unit: participants]
  no children | 23 | 13 | 36
  one livebirth | 7 | 7 | 14
  two livebirths | 0 | 9 | 9
  three livebirths | 0 | 1 | 1
number of previous cesarean sections [Number; unit: participants]
  none | 22 | 14 | 36
  one | 8 | 8 | 16
  two | 0 | 7 | 7
  three | 0 | 1 | 1
previous vaginal deliveries [Number; unit: participants]
  no vaginal deliveries | 28 | 26 | 54
  previous vaginal deliveries | 2 | 4 | 6
infertility [Number; unit: participants]
  no infertility | 1 | 6 | 7
  primary infertility | 19 | 12 | 31
  secondary infertility | 10 | 12 | 22
duration of infertility [Median (Inter-Quartile Range); unit: years] | 2 [2 to 3] | 3 [2 to 4] | 2.5 [2 to 3]
Dysmenorrhea [Number; unit: participants]
  participants having dysmenorrhea | 27 | 11 | 38
  participants not having dysmenorrhea | 3 | 19 | 22
chronic pelvic pain [Number; unit: participants]
  participants having chronic pelvic pain | 9 | 4 | 13
  participants not having chronic pelvic pain | 21 | 26 | 47
Dyspareunia [Number; unit: participants]
  participants having dyspareunia | 12 | 3 | 15
  participants not having dyspareunia | 18 | 27 | 45
Menorrhagia [Number; unit: participants]
  participants having menorrhagia | 6 | 3 | 9
  participants not having menorrhagia | 24 | 27 | 51
categorization of participants according to body mass index [Number; unit: participants]
  lean | 16 | 3 | 19
  overweight | 13 | 13 | 26
  obese | 1 | 14 | 15

OUTCOME MEASURES:

1. Primary Outcome: Serum Nesfatin 1
Description: Venous samples for measurement of nesfatin-1 were taken by venipuncture from patients during the laparoscopy procedure immediately after initial evaluation and before any intervention.The blood samples were centrifuged immediately after their collection at 5000 rpm for 10 min and serum samples were stored at -20 °C until analysis. Nesfatin-1 was measured by Enzyme-Linked Immuno Sorbent Assay "ELISA" technique using commercially available kits (Boster Biological Technology Human Nesfatin-1 ELISA kits, Catalog number EK1138, USA) in the Central Labs of Ain Shams University Hospitals.
Time Frame: 24 hours
Population: In the endometriosis group, two patients were stage I, one was stage II, 12 were stage III and 15 were stage IV according to the revised ASRM scoring system. In the control group, 13 had polycystic varies, 11 had variable pelvic peritoneal adhesions, 4 had tubal block , one had unilateral ovarian cyst and one patient had atrophic ovaries.
Measure: Median (Inter-Quartile Range); unit: picogram/millilitre
Arm/Group | Endometriosis | Control
Number analyzed (Participants) | 30 | 30
picogram/millilitre | 190 [150 to 280] | 510 [410 to 600]
Statistical Analysis 1: Comparison: Endometriosis vs Control; Normality of numerical data distribution was examined by the Shapiro-Wilk. Normally distributed numerical variables were presented as mean±SD and inter-group differences were compared using unpaired t test. Skewed numerical variables were presented as median and interquartile range and between-group differences were compared using Mann-Whitney U test. Ordinal data were compared using the chi-squared test for trend. Correlations among numerical variables were tested by Spearman rank correlation; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: All participants were followed up in the hospital for 48 hours and then contacted by phone for another one week till surgical sutures were removed. Then, they were followed by phone for another one month for any adverse events.
Arm/Group | Endometriosis | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No